CLINICAL TRIAL: NCT01565629
Title: Computer- Assisted Cognitive-Behavioral Treatment for Anxiety Disorders in Children With Autism Spectrum Disorders
Acronym: CCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCAL-2012
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Autism; Asperger's Syndrome; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder; Obsessive-compulsive Disorder
Keywords: Autism; Asperger's Syndrome; Treatment; Cognitive-behavioral therapy; Anxiety; Children; Therapy
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist Condition (No Intervention): Children in this condition will withhold from any type of intervention for a period of 12 weeks.
- Computer Assisted CBT (Experimental): Those who choose to participate will be required to attend 4 assessments - pre-treatment (week 0), mid-treatment (week 8), post-treatment, and a 4th assessment for a 3 month Follow-up. All children regardless of condition will follow the CCBT protocol (Camp Cope-A-lot), which is the computer-assisted intervention being examined in this study. The first 6 levels of this program are skill building levels to be completed by the user. The remaining 6 levels are completed with the therapist and consist of exposure tasks and rehearsal geared toward each child.
  Interventions: Behavioral: Computer assisted cognitive behavioral therapy.

INTERVENTIONS:
Behavioral: Computer assisted cognitive behavioral therapy. — Those who choose to participate will be required to attend 4 assessments - pre-treatment (week 0), mid-treatment (week 8), post-treatment, and a 4th assessment for a 3 month Follow-up. All children regardless of condition will follow the CCBT protocol (Camp Cope-A-lot), which is the computer-assisted intervention being examined in this study. The first 6 levels of this program are skill building levels to be completed by the user. The remaining 6 levels are completed with the therapist and consist of exposure tasks and rehearsal geared toward each child.
  Other Names: CCAL; CCBT; Camp Cope-A-Lot
  Arms: Computer Assisted CBT

SUMMARY:
This study will examine the efficacy of a computerized cognitive behavioral therapy (CCBT) program for children with anxiety and autism spectrum disorders.

DETAILED DESCRIPTION:
Many children who have an autism spectrum disorder (ASD) experience substantial anxiety that can cause impairment above that of an ASD alone. Few studies have examined effective treatment options for anxiety in this population.Preliminary studies have established the efficacy of computer-assisted cognitive behavioral therapy in otherwise typically developing youth with anxiety. Accordingly, this study seeks to examine the efficacy of computer assisted CBT in children with autism and ASD. A randomized-control trial will examine the ability of computer-assisted CBT to treat anxiety in comparison to a waitlist condition. This study will recruit approximately 40 youth ages 7-12 years. Significant reductions in anxiety severity and overall improvement of functioning will establish this treatment's ability to treat anxiety. This study aims to evaluate the acute efficacy of CCBT relative to WAITLIST in children with ASD and comorbid anxiety disorders;examine the short-term durability of treatment gains for youth receiving CCBT; examine whether, relative to WAITLIST, CCBT results in improved social; adaptive; and global functioning, as well as reduced child- and parent-rated anxiety symptoms; and examine whether, relative to WAITLIST, CCBT is associated with greater satisfaction and consumer acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient children with an autism spectrum disorder (see #2 below) between the ages 7-12 years.
2. Meets criteria for a diagnosis of an autism spectrum disorder using scores from the Autism Diagnostic Observation Schedule and Childhood Autism Rating Scale-II High Functioning Version.
3. Meets DSM-IV criteria for a diagnosis of one of the following anxiety disorders: separation anxiety disorder (SAD), generalized anxiety disorder (GAD), social phobia, panic disorder or specific phobia as determined by the ADIS-IV-C/P (with CSR 4) and all available information.
4. Minimum score of 12 on the PARS Severity Scale
5. Child has a Full Scale and Verbal Comprehension IQ > 85 as assessed on the KBIT-2.
6. Subjects with co-morbid depression, ADHD, tic disorder or disruptive behavior disorders will be acceptable as long as the anxiety disorder is primary (i.e., most impairing/distressing).

Exclusion Criteria:

1. Receiving concurrent psychotherapy, social skills training, or behavioral interventions (e.g., applied behavior analysis). Families will have the option of discontinuing such services to enroll in the study.
2. New Treatments: Initiation of an antidepressant within 10 weeks before study enrollment or an antipsychotic 6 weeks before study enrollment. No new alternative medications, nutritionals or therapeutic diets within 8 weeks of study enrollment.
3. Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxiolytics) within 6 weeks before study enrollment, or any change in alternative medications that might have behavioral effects within 4 weeks prior to the study baseline assessment.
4. (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.
5. Lifetime DSM-IV bipolar, schizophrenia or schizoaffective disorders; or Substance abuse in past 6 months.
6. Unwillingness of parents to make the commitment to accompany their child for multiple study visits.
7. Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study or if the computer-assisted CBT is not a good avenue of treatment for the child.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale | After an average of 12 weeks (Post-treatment)

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule: Parent and Child Versions | After an average of 12 weeks (Post-treatment)
Clinical Global Impression - Severity Scale | After an average of 12 weeks (Post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Storch, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, St. Petersburg, Florida, United States